CLINICAL TRIAL: NCT04943536
Title: Bicalutamide Implants (Biolen) With Radiation Therapy in Patients With Localized Prostate Cancer
Acronym: BiolenRT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alessa Therapeutics Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-002; ZIABC010850 (NIH); ZIABC011552 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — bicalutamide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biolen+Radiation Therapy (Experimental): Localized single delivery of the Biolen implant (polymer + bicalutamide) with radiation therapy
  Interventions: Drug: bicalutamide; Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Drug: bicalutamide — localized anti-androgen therapy
Radiation: Stereotactic body radiation therapy — localized radiation therapy

SUMMARY:
This study will be undertaken to evaluate the feasibility of replacing systemic Androgen Deprivation Therapy (ADT) with targeted local delivery of an anti-androgen agent alone in patients in whom ADT + radiation therapy is indicated for the treatment of localized prostate cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm feasibility study. Up to 20 participants will be recruited to assess the safety and patient tolerance of Biolen for the localized delivery of bicalutamide into the prostate when delivered with radiotherapy.

At baseline, patients will undergo multiparametric MRI of the prostate. Study participants will have placement of the drug eluting Biolen implants. At the 8 week timepoint, participants will undergo repeat multiparametric MRI.

Participants will receive standard of care radiation therapy on weeks 9-11 and will be followed through 2 years post radiation. A third and fourth multiparametric MRI will be performed at 6 and 24 months after completion of radiation. Clinical labs and correlative sample collection and patient quality of life questionnaires will be administered at follow-up visits. Following completion of follow-up or removal from protocol, patients may be offered enrollment on long-term follow up protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven localized prostate cancer in whom prostate radiation and ADT is appropriate therapy (such as Intermediate Risk localized prostate cancer)
* Patients must have at least 1 MRI detected; biopsy proven prostate cancer.
* Patients diagnosed as one of the following:

  1. National Comprehensive Cancer Network (NCCN) intermediate risk prostate cancer, OR
  2. NCCN high risk prostate cancer due to Gleason Grade 4 or 5 AND refuses to receive systemic ADT, OR
  3. NCCN high risk prostate cancer due to Prostate Specific Antigen (PSA) > 20 AND refuses to receive systemic ADT.
* Age >18 years.

Exclusion Criteria:

* NCCN high risk patients eligible for treatment with systemic ADT who do not refuse systemic ADT.
* Patients receiving prior radiotherapy or surgery for prostate cancer.
* Patients receiving prior or ongoing ADT.
* Study participant unwilling or unable to undergo MRI, including patients with contra-indications to MRI, such as cardiac pacemakers, non-compatible intracranial vascular clips, etc.
* Use of 5 alpha reductase inhibitors (e.g. Finasteride or Dutasteride) within 3 months of screening or total use within the last two years prior to screening of > 3 months.
* Prostate volume more than 80 cc at prior MRI imaging.
* International Prostate Symptom Score ≥ 20.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of replacing systemic androgen tx with targeted local delivery | 27 months
  Ability to successfully implant the prostate with Biolen and a lack of implant toxicity that interferes with the capacity to complete intended radiation therapy.

SECONDARY OUTCOMES:
Adverse Events | through 27 months
  toxicity of localized delivery of bicalutamide
MRI changes | baseline versus 8 weeks post biolen implantation and 6 months post RT
  prostate and tumor volume changes
Biochemical progression free survival | 24 months post RT
  rate of biochemical progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Citrin, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No